CLINICAL TRIAL: NCT02856945
Title: Clinical Criteria for Decision Support Regarding Emergency Radiography for Knee Acute Traumatism in Order to Identify Bone Fracture Among Children.
Brief Title: Knee Injury Decision
Acronym: KID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0518
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Bone Fracture; Knee Trauma
Keywords: fracture; children; knee; clinical criteria; decision making
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
At this time, there is no standardization for knee trauma care in children. Each physician is free to resort or not to radiography to verify or dispel bone fracture, depending on radiographic device availability. This decision is based on trauma severity, clinical features, and physician experience.

Knee traumatisms are a common reason of consultation. In emergency departments, radiographic use is widespread for those traumatisms, but not in private practice.

Most of those knee traumatisms includes soft tissue lesion, for which radiography gives no details. Yet, radiography exposes bone fracture which may require a specific orthopaedic care. Then, it seems beneficial to highlight simple and reproducible clinical criteria in order to identify severe knee traumatisms, requiring radiography to assess bone fracture.

Those criteria should have a sensibility close to 1, and the highest specificity. Such criteria could significantly decrease the number of radiography thus irradiation, emergencies waiting time, and consultation expenses without missing bone fracture.

Ottawa knee rules for adults are: age 55 years older, tenderness at head of fibula, isolated tenderness of patella inability to flex to 90°, inability to bear weight on 4 steps both immediately and in the emergency department. Presence of one of those criteria required front and profile radiography to assess bone fracture.

However, few studies have been conducted among children, and they do not confirm the use of those criteria targeting fracture screening. Data are contradictory and they do not allow concluding that such criteria could be of benefit for children. Moreover, studies only consider adults clinical criteria. This study would be the first to implement specific paediatric criteria, which make this study original.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 1 to 17 years old included
* Knee traumatism (distal third of femur and proximal third of tibia/fibula)
* Traumatism not older than 7 days

Exclusion Criteria:

* Isolated knee wound
* Loss of awareness
* Paraplegia

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Knee traumatism at HFME hospital
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
clinical criteria sensitivity | when radiography results are available (day 1)
  sensitivity will be evaluated for each clinical criterion, with the radiographic gold standard. Sensitivity will be compared by Mc Nemar paired test, or by Fischer exact test if Mc Nemar test conditions are not fulfilled.

SECONDARY OUTCOMES:
criteria specificity | when radiography results are available, at inclusion day (day 1)
  specificity will be evaluated for each clinical criterion, with the radiographic gold standard. Specificity will be compared by Mc Nemar paired test, or by Fischer exact test if Mc Nemar test conditions are not fulfilled
Positive and negative predictive values | when radiography results are available, at inclusion day (day 1)
Radiographic use reduction | when radiography use is determined
  The number of radiographic use will be measure to identify any variation in this procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Karine CORREARD, MD, Principal Investigator — Hospices Civils de Lyon, HFME
Locations (1):
- Hospices Civils de Lyon, HFME. 32 Avenue Doyen Jean Lépine, Bron, France